CLINICAL TRIAL: NCT05776550
Title: A Prospective Registry to Assess the Safety and Efficacy of Distal Radial Approach (SAFE-BOX)
Brief Title: Safety and Efficacy of Distal Radial Approach (SAFE-BOX)
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Other Study IDs: 9-2021-0048
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Safety; Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Prospective Registry to assess the Safety and Efficacy of Distal Radial Approach

DETAILED DESCRIPTION:
Anaphylactic radial approach is now recognized as a basic technique in coronary artery procedures. The main advantage is increased stability due to the reduction of massive bleeding and increased patient comfort because it can move immediately after the procedure. The operator prefers access to the right radial artery because of the comfort of performing the procedure on the right side of the patient. However, the operator should frequently replace it with a left radial artery approach for various reasons, including 1) closure of the right radial artery, 2) difficulty accessing the coronary artery due to severe gambling of the radial artery, and 3) hemodialysis of the right radial artery.

As for prognosis, the left and right radial artery approaches are similar. However, the left radial artery approach is bound to experience anthropological discomfort in which the operator has to lean toward the patient. An easy solution is the approach from the anatomical left snuff box located on the back of the hand to the distal radial artery. Recently, the left snuffbox approach has been reported, and attempts are increasing in many countries. However, it is true that there is still a difference in diameter of the radial artery through the distant radial artery approach and concerns about percutaneous coronary intervention through this compared to the classical radial artery approach. Recent studies have published studies on the stability and effectiveness of distant radial artery approaches, but they are still small, and studies on specific subgroups are very scarce. Furthermore, data on the current status and performance in Korea so far is very scarce. Therefore, through this study, we would like to systematically collect and analyze data on the status and performance of the approach through the distant radial artery approach to find out the stability and effectiveness of various patient groups, treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 20 years of age
2. Patients requiring coronary angiography or intervention
3. Patients with palpable distant radial artery

Exclusion Criteria:

1. Patients with distant radial artery too small or not palpable
2. Pregnant women
3. Patients not appropriate for the researcher to judge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Evaluate the success rate of coronary angiography and intervention in patients with palpable radial artery
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Success rate of examination and procedure | through procedure completion, up to 24 hours
  Success rate of examination and procedure

SECONDARY OUTCOMES:
the success rate of the puncture | through procedure completion, up to 24 hours
  the success rate of the puncture
puncture time | through procedure completion, up to 24 hours
  puncture time
complications of the puncture region | the first outpatient visit after discharge
  complications of the puncture region

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Study Director — Severance Hospital
Locations (1):
- Yongcheol Kim, Yongin, Gyeonggi-do, South Korea